CLINICAL TRIAL: NCT02702206
Title: Effect of Ultrasound-guided Hyaluronic or Corticosteroid Injections in Patients With Chronic Subacromial Bursitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20131202R; MOST 103-2314-B-341 -003 -MY2 (Other Grant/Funding Number: Ministry of Science and Technology)
Record Dates: First submitted 2014-11-18; First posted 2016-03-08 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2017-01

CONDITIONS: Shoulder Pain; Subdeltoid Bursitis; Subacromial Bursitis
Keywords: Shoulder pain; subdeltoid bursitis; subacromial bursitis; intra-bursa injection
MeSH Terms: conditions — Shoulder Pain | interventions — Adrenal Cortex Hormones; Triamcinolone; Hyaluronic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- corticosteroids SASD injection (Experimental): under US guidance 2ml triamcinolone (1ml/10mg), 0.5ml distilled water and 1ml 1% lidocaine
  Interventions: Drug: corticosteroids
- hyaluronic acid (ARTZ) SASD injection (Experimental): under US guidance 2.5ml HA (ARTZ, 1% sodium hyaluronate solution, 10mg/mL, molecular weight 0.9x106Da) and 1ml 1% lidocaine
  Interventions: Drug: hyaluronic acid
- normal saline SASD injection (Placebo Comparator): under US guidance 2.5ml normal saline and 0.5ml distilled water and 1ml 1% lidocaine
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: corticosteroids — under US guidance, 2ml triamcinolone (1ml/10mg), 0.5ml distilled water and 1ml 1% lidocaine
  Other Names: triamcinolone
  Arms: corticosteroids SASD injection
Drug: hyaluronic acid — under US guidance, 2.5ml HA (ARTZ, 1% sodium hyaluronate solution, 10mg/mL, molecular weight 0.9x106Da) and 1ml 1% lidocaine
  Other Names: ARTZ
  Arms: hyaluronic acid (ARTZ) SASD injection
Drug: normal saline — under US guidance, 2.5ml normal saline (placebo group). 0.5ml distilled water and 1ml 1% lidocaine
  Other Names: placebo group
  Arms: normal saline SASD injection

SUMMARY:
A randomized controlled trial to compare the effect of ultrasound-guided hyaluronic or corticosteroid injections in patients with chronic subacromial bursitis.

DETAILED DESCRIPTION:
Chronic subacromial bursitis (SAB) is a common shoulder disorder characterized by chronic shoulder pain with a painful arc of motion, which commonly occurs during abduction and sometimes during internal rotation of the shoulder. In addition, the extremes of all passive movements are painful. The range of motion (ROM) of the shoulder is usually not limited or is limited in a non-capsular pattern (mainly abduction and internal rotation). All resisted movements are painless or equally painful, and there is also tenderness over the deltoid region. The diagnosis of SAB remains doubtful until it is confirmed by an infiltration with local anesthetic.

The injections can be performed by palpation (using anatomical landmarks to place the needle) or with ultrasound (US) guidance (with visualization of the needle tip at the target location). The chief advantage of an ultrasound-guided intervention is the ability to use real-time, dynamic imaging without ionizing radiation. Previous studies have demonstrated that ultrasound-guided injection ensures correct needle placement and delivery of the medicine to the target, and improved clinical outcomes with ultrasound-guided subacromial-subdeltoid (SASD) corticosteroid injections.

Although SASD corticosteroid injections has been proven effective in treatment of chronic subacromial bursitis, in clinical practice, some patients fear the side effects of the corticosteroids. In the last few years, hyaluronic acid (HA) injection has been used for treatment of different kinds of shoulder disorders, including subacromial impingement syndrome, frozen shoulder, and rotator cuff tears, with variable results. However, treatment of chronic SAB with hyaluronic acid has never been reported before. Besides, some authors used combination of normal saline and lidocain as the placebo, which might not be a true placebo because lidocain can be an active medicine. Therefore, the purpose of this study is to compare the effectiveness of SASD corticosteroid, HA, and normal saline injection in treatment of patients with chronic SAB.

ELIGIBILITY:
Inclusion Criteria:

1. shoulder pain for more than 1 month
2. age ≥ 20 years old
3. painful abduction or internal rotation with a visual analog scale (VAS) pain score ≥4
4. the presence of a painful arc of motion or pain at the middle to terminal range of shoulder abduction or internal rotation with a soft end feel
5. tenderness over the subacromial bursa
6. a reduction in pain of ≥40% on active shoulder abduction or internal rotation at the terminal range after injection of 3ml of 1%lidocain into the SASD bursa under ultrasound (US) guidance.

Exclusion Criteria:

1. a history of uncontrolled chronic diseases, e.g., malignant neoplasms, blood dyscrasia, and infection
2. previous surgery of the affected shoulder
3. any evidence of a rotator cuff tear or tendinopathy, demonstrated by positive resistive tests or sonographic findings
4. calcification of the rotator cuff, demonstrated by x-ray or sonographic findings
5. the presence of arthritis, such as inflammatory arthritis (e.g., rheumatoid arthritis, seronegative spondyloarthropathy, or crystal-related arthropathy), osteoarthritis, frozen shoulder, subacromial spurs, or deformity of the acromion
6. the presence of instability of the affected shoulder
7. a previous fracture near the shoulder region
8. the presence of cervical radiculopathy or myelopathy
9. having received a corticosteroid or hyaluronic acid subacromial or shoulder joint injection in the past 3 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2014-08; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline VAS pain score | baseline and 2 weeks
  The VAS scores for pain were obtained using a 100-mm-long horizontal line, with 0 mm on the left indicating no pain and 100 mm on the right indicating very severe pain.

SECONDARY OUTCOMES:
the active ROM | between these time points: baseline, 2 weeks, 4 weeks (end of the intervention), 8 weeks, and 16 weeks
  The maximal active ROMs of the affected shoulder will be measured using a goniometer under the guidelines of the American Academy of Orthopedic Surgeons. These measurements included abduction in the frontal plane, forward flexion, internal rotation, and external rotation with the arm at 0 degrees of abduction.
Change of scores of the Shoulder Pain and Disability Index (SPADI) | between these time points: baseline, 2 weeks, 4 weeks (end of the intervention), 8 weeks, and 16 weeks
  The total SPADI score, which ranges between 0 and 100, is calculated by averaging the scores from the pain and disabilities subclasses.
Change of the Shoulder Disability Questionnaire (SDQ) | between these time points: baseline, 2 weeks, 4 weeks (end of the intervention), 8 weeks, and 16 weeks
  The SDQ is a symptoms-related questionnaire containing 16 items describing common situations that may induce symptoms in patients with shoulder disorders. By responding 'yes', 'no', or 'not applicable', the final score is obtained by dividing the number of positively scored items by the total number of applicable items and then multiplying this number by 100, which results in a final score ranging between 0 (no disability) and 100 (the worst situation).
Change of 36-item Short-Form Health Survey (SF-36) | between these time points: baseline, 2 weeks, 4 weeks (end of the intervention), 8 weeks, and 16 weeks
  The SF-36 is a 36-item questionnaire that evaluates the quality of life. It is composed of 8 subscales: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Each subscale has a score range of 0 to 100, with a higher score indicating better health status.Patient's evaluation of the treatment effect. Patient's evaluation of the treatment effect consists of the answer to one question: "Is the treatment effective?" scored on a Likert scale (very effective=1, effective=2, not effective=3, worse=4, much worse=5).

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Fen Hsieh, M.D, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Hsieh LF, Lin YJ, Hsu WC, Kuo YC, Liu YC, Chiang YP, Wang CP. Comparison of the corticosteroid injection and hyaluronate in the treatment of chronic subacromial bursitis: A randomized controlled trial. Clin Rehabil. 2021 Sep;35(9):1305-1316. doi: 10.1177/02692155211007799. Epub 2021 Apr 15. PMID 33858205